CLINICAL TRIAL: NCT04045262
Title: Clinical Validation of Continuous and Non-invasive Monitoring of Effective Pulmonary Volume Based on Exhaled CO2 Kinetics in Ventilated Patients.
Brief Title: Clinical Validation of Continuous and Non-invasive Monitoring of Effective Pulmonary Volume.
Status: Completed | Type: Observational
Sponsor: Fernando Suarez Sipmann (Other)
Responsible Party: Sponsor-Investigator, Fernando Suarez Sipmann, MD PhD Intesive Care Medicine, Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Organization: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Other Study IDs: EELVC02
Record Dates: First submitted 2019-08-02; First posted 2019-08-05 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to evaluate/validate a new non-invasive method to continuously monitor effective lung volume in critically ill patients.

DETAILED DESCRIPTION:
The capnodinamyc method is a new monitoring method that provides continuous (breath by breath) measurements of effective pulmonary blood flow (EPBF) and effective end-expiratory l lung volume (EELVCO2). The former refers to the non-shunted fraction of cardiac output and the latter to the functional end-expiratory lung volume (EELV) that contains CO2.

The capnodynamic method is based on the advanced analysis of CO2 kinetics and the law of Conservation of mass. It states that lungs have to eliminate a similar amounts of CO2 as produced by aerobic metabolism and reaches the lung via pulmonary perfusion. For its calculation, two different measurements are needed:

1. Exhaled CO2 measured by infrared optic sensor technology placed in a mainstream configuration between the endotracheal tube and the "Y" piece of the ventilator respiratory circuit.
2. Flow, airway pressure and ventilatory volumes measured by the mechanical ventilator spirometer.

The method requires the generation of cyclic small changes in the alveolar concentration of CO2 which is achieved by introducing a slightly modified breathing pattern. It consists of adding a short expiratory hold in each 3 out of 9 consecutive breaths and requires the patient to be in passive breathing conditions under mechanical ventilation.

EPBF and EELVCO2 have been validated in experimental conditions and the first validations in patients in the setting of general anesthesia are under way.

Methods:

This study on EELVCO2 in critically ill patients involves 2 types of evaluations:

The validation of absolute values of EELV by comparing it with CTsan. The trending ability of EELVCO2 in critically ill patients by comparing it with EIT.

A calculated sample size of 30 patients is required for each objective.

ELIGIBILITY:
Inclusion Criteria:

* All patients on mechanical ventilation in passive breathing conditions in which a thoracic CTscan has been indicated for medical reasons and those with an EIT and a continuous cardiac monitoring
* Informed consent

Exclusion Criteria:

* Hemodynamic instability
* Presence of barotrauma/ pneumothorax
* Presence of bronchopleural fistulas
* Thorax alterations that preclude the positioning of the EIT electrode belt (usually at the IV intercostal space).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients undergoing mechanical ventilation
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Validation of the measurement of absolute values of effective lung volume | 1 day
  To validate the measurement of absolute values of effective lung volume by the capnodynamic method previously described, as an estimate of end-expiratory lung volume. For this purpose the capnodynamic method will be compared with gold standard reference method for measuring lung volumes, the computerized tomography scan (CTscan).
Analyze to which pulmonary compartments does effective lung volume most closely correlate | 1 day
  Tomographic aeration level according to the density distribution analysis (non aerated, poorly aerated, normally and hyper aerated) does effective lung volume most closely correlate; taking into account that the CTscan measures an anatomic rather than a functional lung volume.
Improvement of capnodynamic ELV measurement | 1 day
  To determine the effects of lung collapse on the accuracy and precision of the capnodynamic ELV measurement.
Trending ability of the capnodynamic end-expiratory lung volume method | 1 day
  Breath by breath changes in EELVCO2 will be compared with breath by breath changes in lung aeration measured by electrical impedance tomography.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Suarez Sipmann, MD PhD, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de la Princesa, Madrid, Spain

REFERENCES:
- [Derived] Sanchez Giralt JA, Tusman G, Wallin M, Hallback M, Perez Lucendo A, Sanchez Galindo M, Abad Santamaria B, Paz Calzada E, Garcia Garcia P, Rodriguez Huerta D, Canabal Berlanga A, Suarez-Sipmann F. Clinical validation of a capnodynamic method for measuring end-expiratory lung volume in critically ill patients. Crit Care. 2024 Apr 30;28(1):142. doi: 10.1186/s13054-024-04928-w. PMID 38689313